CLINICAL TRIAL: NCT00299065
Title: Assessment of Safety, Tolerability, and Pharmacokinetics of Zileuton Injection in Patients With Asthma
Brief Title: Safety Study of Zileuton Injection in Patients With Asthma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Critical Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTI-04-C05-201
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Asthma
Keywords: Asthma, bronchial; Asthma, exercise-induced; Anti-asthmatic agents
MeSH Terms: conditions — Asthma; Asthma, Exercise-Induced | interventions — zileuton

INTERVENTIONS:
Drug: Zileuton injection

SUMMARY:
The prevalence of asthma continues to increase. Despite the large number of available therapies, many patients continue to require emergency deparment (ED) visits and intensive therapy. However, ED visits continue to be a major contributor to the healthcare cost of asthma treatment. In the United States alone, asthma is the 11th most common reason for ED visits, with ED visits and hospitalizations accounting for almost 50% of the healthcare cost for asthma. Additionally, while only 20% of asthmatics have had ED visits or hospitalizations, these patients account for over 80% of the direct costs for asthma treatment. Current National Asthma Education and Prevention Program (NAEPP) guidelines regarding management of acute asthma exacerbations in the ED setting include: oxygenation for most patients, inhaled short-acting β2-agonists and systemic corticosteroids.

Zileuton, a specific 5-lipoxygenase inhibitor, has been extensively studied in inflammatory diseases such as asthma, which involve leukotrienes as mediators of inflammation. Zileuton Immediate Release (IR) tablets (Zyflo®) were approved by the Food and Drug Administration (FDA) in December 1996 for the prevention and treatment of asthma in adults and children 12 years of age and older. The results of the 2 pivotal studies in asthmatics with zileuton IR tablets demonstrated that zileuton at a dose of 600 mg QID produced and maintained a lasting improvement of lung function. In addition to the lasting effect of zileuton, an acute bronchodilation (as early as 60 minutes) was observed after administration of the first 600 mg oral dose.

This acute bronchodilator effect may benefit patients during an acute exacerbation of asthma when added to the usual care in the ED or clinic setting. Critical Therapeutics has developed an injectable formulation of zileuton that will be explored for use in acute asthma exacerbations. This initial study is intended to provide PK data, information on safety and tolerability and some indication of pharmacologic activity as evidenced by lung function changes. In an attempt to enhance the potential for observing effects on lung function, only those patients with a demonstrated ability to respond by an increase in FEV1 of at least 10% within 3 hours after oral zileuton dosing will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Morning FEV1 of 40-80% of predicted normal
* Evidence post-bronchodilator increase in FEV1 of at least 15%
* Evidence of at least 10% increase in FEV1 within 3 hours after oral 600 mg zileuton dose
* Signed IRB approved informed consent
* Patients must be willing and able to withhold:
* short acting β2-agonists for at least 6 hours prior to spirometry
* inhaled corticosteroids (ICS) for at least 24 hours prior to sprirometry
* long acting β2-agonists (LABA) for 7 days and be willing and able to switch from a LABA/ICS combination product to a monotherapy ICS product

Exclusion Criteria:

* Females of childbearing potential not using effective contracception
* Any uncontrolled systemic disease other than asthma
* Patient with known hypersensitivity to zileuton IR tablets or zileuton injection or any of the components found therein
* An upper or lower respiratory tract infection within 2 weeks of screening
* An ED visit or hospitalization for asthma within 3 months of screening
* Oral or parenteral corticosteroid use for asthma exacerbation within 3 months of screening
* Current cigarette smoker and/or >10 pack-year smoking history
* History of hepatitis B (HBV) or hepatitis C infection or other active liver disease or chronic hepatitis
* Screening ALT >1.5x ULN
* Patient with impaired renal function or serum creatinine >1.5x ULN
* History of HIV infection
* History of drug or alcohol abuse within 1 year of screening
* Patient taking any of the following asthma/allergy medications:
* Anti-IgE meds within 3 months of screening
* Zileuton IR tablets within 1 month of screening
* Inhaled or oral steroids not stable for at least 1 month
* Theophylline, cromolyn, or nedocromil within 7 days of screening
* Leukotriene receptor agonists within 7 days of screening
* Warfarin, propranolol, inhaled or sytemic anticholinergics within 7 days of screening
* Long acting beta agonist within 7 days of screening
* Oral beta-2 agonists within 12 hours of screening
* Immunotherapy injections not in a stable dosing phase
* Female patient who is pregnant or breast-feeding or plans to become pregnant during the study period
* Participation in another research study within 30 days of screening
* Patient is the Investigator or other staff or relative who is directly involved in the conduct of the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2006-01; Study Completion 2006-06

PRIMARY OUTCOMES:
Clinical laboratory tests through 48 hours post-injection
Vital signs through 10 hours post-injection
Pulse oximetry through 10 hours post-injection
Injection site evaluations through 10 hours post-injection
Adverse event assessments through 48 hours post-injection
Blood samples for PK through 10 hours post-injection

SECONDARY OUTCOMES:
Spirometry through 10 hours post-injection
Peak expiratory flow rates through 20 min. post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Dana Hilt, MD, Study Director — Critical Therapeutics Incorporated
Locations (10):
- United States (10):
  - Allergy & Asthma Specialist Medical Group, Huntington Beach, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Colorado Allergy and Asthma Centers, PC, Englewood, Colorado
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Clinical Research Center, L.L.C., St Louis, Missouri
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy Associates Research Center, Portland, Oregon
  - Western Sky Medical Research, El Paso, Texas

REFERENCES:
- [Background] Fuhlbrigge AL, Adams RJ, Guilbert TW, Grant E, Lozano P, Janson SL, Martinez F, Weiss KB, Weiss ST. The burden of asthma in the United States: level and distribution are dependent on interpretation of the national asthma education and prevention program guidelines. Am J Respir Crit Care Med. 2002 Oct 15;166(8):1044-9. doi: 10.1164/rccm.2107057. PMID 12379546
- [Background] Colice GL, Burgt JV, Song J, Stampone P, Thompson PJ. Categorizing asthma severity. Am J Respir Crit Care Med. 1999 Dec;160(6):1962-7. doi: 10.1164/ajrccm.160.6.9902112. PMID 10588614
- [Background] Rodrigo GJ, Rodrigo C, Hall JB. Acute asthma in adults: a review. Chest. 2004 Mar;125(3):1081-102. doi: 10.1378/chest.125.3.1081. PMID 15006973